CLINICAL TRIAL: NCT01985269
Title: Modified Directly Observed Antiretroviral Therapy (M-DART): An Intensive, Nurse-directed, Home-centered, Treatment Strategy to Reduce Mortality and Loss to Follow-up in High-risk HIV-infected Patients Initiating Antiretroviral Therapy
Brief Title: Modified Directly Observed Antiretroviral Therapy
Acronym: M-DART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Moi University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, ABRAHAM M. SIIKA, MBChB, MMed, MS, Associate Professor of Medicine, Moi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AID-623-A-00-08-00003
Record Dates: First submitted 2013-10-24; First posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: HIV
Keywords: High risk; ART naive
MeSH Terms: interventions — House Calls

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home visits (Active Comparator): Minimal physical examination at home Drug adherence/pill counts
  Interventions: Other: Home visits
- Control (No Intervention): Normal standard of care

INTERVENTIONS:
Other: Home visits — The participants' vital signs (blood pressure, temperature, pulse rate, respiratory rate, and arterial oxygen saturation) will be taken and a limited physical examination (e.g. oral cavity for thrush, Kaposi's lesions, ulcers and dehydration; skin for rash, herpes zoster and dehydration; eyes for jaundice and pallor, gross neurological function such as ability to walk without difficulty, presence of facial droop, one-sided body weakness etc.) conducted. The nurse will then review medications adherence before observing the study participant swallow their pills (antiretrovirals, anti-TB, antibiotics, and analgesics).
  Other Names: Treatment arm; Intervention arm
  Arms: Home visits

SUMMARY:
M-DART Study is a randomized clinical trial comparing the effectiveness of a home-based modified directly observed antiretroviral (ART) treatment strategy to clinic-based standard of care in patients with HIV/AIDS in Port Victoria, Busia, Kitale, Chulaimbo and Khunyangu, Kenya.

Hypothesis 1a: It is feasible to implement M-DART in remote, poverty stricken, high-HIV prevalence rural communities in western Kenya.

Hypothesis 1b: M-DART will be a more effective strategy than standard of care (High-Risk Express Care) in reducing mortality and LTFU in patients at the highest risk of dying following ART initiation.

Hypothesis 2: M-DART will be cost effective over the 48-week study period

Hypothesis 3a: Patients enrolled in M-DART will have higher quality of life scores at 24 and 48 weeks as compared to the control patients.

Hypothesis 3b: Patients enrolled in M-DART will have lower HIV related stigma scores at 24 and 48-weeks as compared to the control patients.

DETAILED DESCRIPTION:
Mortality and lost to follow-up (LTFU) rates amongst adult African HIV-infected patients on antiretroviral therapy (ART) are high, especially so in the first 12 months of treatment. Although the risk factors for death and LTFU in these patients have been elucidated, specific care interventions to reduce both death and LTFU have not been reported. Therefore, there is an urgent need for evidence-based knowledge of care interventions that reduce early mortality and LTFU in HIV-infected patients on ART in sub-Saharan Africa. By informing decision-making processes on resource allocation, treatment and care emphasis-areas and planned strategies, such knowledge would provide treatment programs a great opportunity to lower HIV-related mortality while increasing the benefits of ART.

The USAID-AMPATH Partnership (AMPATH) has enrolled >118,000 HIV-infected patients across 60 urban and rural care sites in western Kenya, >65,000 of whom have initiated ART. To date, >9,000 patients have been confirmed dead, half of whom were on ART. Many more are LTFU, unknown whether they are still alive or not. AMPATH is uniquely placed to perform care intervention trials targeting reduction in mortality and LTFU because:

1. There are sufficient study subjects;
2. It has a protocol-driven care program that will enable the establishment of a control group that is cared for in a standard fashion;
3. The AMPATH Medical Record System (AMRS), a fully computerized system containing >80 million observations collected prospectively for >3.0 million visits will provide easy data storage and retrieval;
4. Experienced investigators from the Moi and Indiana University Schools of Medicine and the World Bank will ensure that the study is executed within acceptable clinical trial standards and in a timely fashion; and
5. It has effective community outreach programs which will increase the chances of the study's acceptability in the community, hence its success.

We propose to perform a randomized clinical trial that will compare the effectiveness of a home-based modified directly observed ART treatment strategy to clinic-based standard of care in reducing both mortality and LTFU soon after ART is initiated. A similar cadre of clinicians will be used for home-based as for clinic-based care in order to enhance comparability of outcomes. A cost effectiveness analysis of the intervention will be performed. The patients' quality of life and perceived HIV stigma will be assessed at study enrollment, 24 and 48 weeks. We will perform the study in two of the remotest AMPATH care sites that have very high HIV-prevalence in the hope that the study's results, if positive, will impact care in communities that need it the most.

2. Specific Aims High mortality and LTFU rates soon after HIV-infected patients initiate ART are two major challenges facing HIV treatment and care programs in sub-Saharan Africa. In the first year of ART, mortality in African patients is as high as 26% despite appropriate treatment. The majority of these deaths occur in the first six months. This mortality rate is 5 - 8 times higher than for similar patients in the developed world. The risk factors for mortality in African patients initiating ART have been well elucidated. These risk factors include: late patient presentation with severe immune degradation and clinically advanced HIV disease; active or latent infections such as tuberculosis, invasive bacterial and fungal; anaemia; malnutrition; care in lower level and fee-for-service centers; male gender; and poor adherence to ART. Similarly, LTFU rates are high. Some care programs have reported LTFU rates as high as 40% in the first 12 months of ART. The risk factors for LTFU have also been reported and some mirror those for death. Recently published data indicate that unreported deaths might be the biggest reason for LTFU. With such abundant knowledge on risk factors for death and LTFU after ART initiation, what is now required is the development, implementation and evaluation of novel treatment and care strategies that target specific risk factors with the aim of mitigating these twin challenges.

The United States Agency for International Development - Academic Model Providing Access to Healthcare (USAID-AMPATH Partnership) is one of the largest public HIV treatment and care programs in sub-Saharan Africa. With care centers in Western, Nyanza and North Rift Valley provinces of Kenya, AMPATH has enrolled over 118,000 HIV-infected patients in 60 urban and rural care sites. Of these patients, >65,000 have initiated ART. To date, more than 9,000 of the >118,000 AMPATH-enrolled HIV-infected patients have been confirmed dead, including more than 5,000 on ART. Current AMPATH's annual LTFU rate is estimated at 8% for patients on ART and 13% for those not on ART. AMPATH's long-term objective is to improve ART outcomes for HIV-infected African patients through the development of replicable, sustainable, cost-effective treatment and care strategies that prevent mortality and prolong survival. Through this proposed research, we would like to study the usefulness of an intensive, nurse-directed, home-centered, modified (three times per week) treatment and follow-up strategy for newly enrolled, HIV-infected, ART-naïve patients at the highest risk of dying after initiating ART. The central hypothesis in this application is that the vast majority of deaths in HIV-infected African patients on ART can be prevented by early identification and aggressive management of HIV- and ART-related complications through close patient monitoring. The rationale behind this proposal is that interventions to interrupt early death in HIV-infected patients on ART are more likely to succeed if HIV and ART-related complications are identified early and appropriate interventions instituted promptly. Furthermore, solutions to HIV care and treatment challenges in sub-Saharan Africa are more likely to be attained if the research conducted addresses the region's specific healthcare needs and the results of such research can be translated into local practice. We plan to accomplish our objective by pursuing the following three specific aims:

1. To develop and implement an intensive, nurse-directed, home-centered, modified directly observed antiretroviral therapy (M-DART) care strategy for high-risk HIV-infected patients initiating ART in remote locations in western Kenya and compare this to the current AMPATH standard of care (High-Risk Express Care).

   * Hypothesis 1a: It is feasible to implement M-DART in remote, poverty stricken, high-HIV prevalence rural communities in western Kenya.
   * Hypothesis 1b: M-DART will be a more effective strategy than standard of care (High-Risk Express Care) in reducing mortality and LTFU in patients at the highest risk of dying following ART initiation.
2. To determine the costs effectiveness of M-DART

   • Hypothesis 2: M-DART will be cost effective over the 48-week study period
3. To determine patients' perception of quality of life and stigma following implementation of M-DART.

   * Hypothesis 3a: Patients enrolled in M-DART will have higher quality of life scores at 24 and 48 weeks as compared to the control patients.
   * Hypothesis 3b: Patients enrolled in M-DART will have lower HIV related stigma scores at 24 and 48-weeks as compared to the control patients.

ELIGIBILITY:
Inclusion Criteria:

Patients who require initiation of ART and fulfill the following AMPATH High-Risk Express Care criteria will be eligible for enrollment into the study.

1. Newly diagnosed HIV-infected patients
2. Age >14 years
3. CD4 count <100 cells/ml
4. ART naïve

Exclusion Criteria:

1. Patients declining home visits
2. Refusal to consent to the study

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Death | 48 weeks
  Death data will be collected at 48 weeks of the study
Lost to follow up | 48 weeks
  Lost to follow up data will be collected at 48 weeks of the study

SECONDARY OUTCOMES:
plasma viral load (pVL) | 48 weeks
  Plasma viral load (pVL) changes at 48 weeks will be measured
CD4 Count (cells/ml) | 48 weeks
  CD4 count changes at 48 weeks will be measured
Weight (Kg) | 48 weeks
  Weight changes at 48 weeks will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Abraham M Siika, MBCHB,MMED,MS, Principal Investigator — Moi University
Locations (1):
- Moi Teaching and Referral Hospital, Eldoret, Rift Valley, Kenya